CLINICAL TRIAL: NCT01628497
Title: Exhaled NO Testing in Filariasis
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Fil-01
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Filariasis
MeSH Terms: conditions — Filariasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive filariasis test: Those testing positive for filariasis
- Filariasis negative

SUMMARY:
This study is looking at the difference in exhaled nitric oxide levels in patients with and without laboratory evidence of filariasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 years or older of either gender
2. Patients presenting with pulmonary symptoms a. Confirmed or suspected asthma patients: i. Patients presenting with symptoms consistent with an acute exacerbation of asthma, including:

1. Wheezing 2. Shortness of breath 3. Chest tightness 4. Cough ii. Disposition to the asthma room after triage and physician evaluation (disposition to other areas of the A&E allowed if due to no available space in the asthma room) iii. Patients are potentially eligible with or without a past history of health care provider diagnosed asthma iv. Patients are potentially eligible regardless of the number of previous episodes of wheezing (i.e. patients with a first episode of bronchospasm are potentially eligible) v. If suspected or documented to have pneumonia or a pulmonary infiltrate, patients are potentially eligible if:

1. They have a dry cough (no production of purulent sputum)
2. They have bronchospasm as manifested by wheezing or need for salbutamol (albuterol) breathing treatments vi. Patients with wheezing are not eligible if they:

1. Have purulent sputum production 2. Have known or suspected:

a. Tuberculosis b. Immunodeficiency c. Congestive heart failure d. Foreign body aspiration b. Patients presenting with a chief complaint of cough: i. Potentially eligible patients will have a cough of greater than one week (seven days) duration ii. Asthma room disposition is not required for these subjects iii. If suspected or documented to have pneumonia or a pulmonary infiltrate, patients are potentially eligible if:

1. They have a dry cough (no production of purulent sputum) iv. Patients with cough are not eligible if:

1. Have purulent sputum production
2. Have known or suspected:

   1. Tuberculosis
   2. Immunodeficiency
   3. Congestive heart failure
   4. Foreign body aspiration
3. Patients will be medically stable at the time of the consent process (see exclusion criteria below)
4. A minimum of 2 years of continuous residence in Guyana at the time of enrollment, exclusive of short trips out of the country (at least 21 of previous 24 months physically in Guyana)
5. English speaking

Exclusion Criteria:

1. Patients less than 6 years of age
2. Patients who do not consent to the study
3. Children (<18 years) without a parent/guardian present
4. Prisoners
5. Patients who appear to be medically or psychologically unstable or felt to be otherwise inappropriate for study enrollment, in the opinion of the investigator or any treating health care provider. This determination will be made on an individual basis, but some of the general criteria to be used in making this determination will be:

   i. The patient appears to be in significant pain ii. The patient appears acutely ill - severe respiratory distress, diaphoretic, altered mental status, active bleeding, actively vomiting, etc.

   iii. Those with respiratory difficulty to the point they cannot speak in complete sentences iv. Chief complaint of sexual assault v. The patient appears acutely intoxicated vi. The patient displays agitated, nervous, restless, or other behavior suggestive of an uncontrolled psychiatric emergency
6. Patients with pulmonary findings felt to be secondary to congestive heart failure, foreign body, bacterial pneumonia, tuberculosis or other clearly defined cause
7. Non-English speaking patients
8. Patients without at least 2 years of residence (exclusive of short trips abroad, total of 21 of 24 previous months physically in Guyana) in Guyana at the time of enrollment

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects:
  * recruited from patients with a chief complaint of wheezing, asthma or cough.
  * assessed by a physician prior to consideration for enrollment into the study
  * screened by the study investigator after evaluation by the physician
  Control subjects:
  Controls will be matched with cases by gender, age and region of residence. They will have non-emergent complaints without respiratory symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown Public Hospital Corporation, Georgetown, Demerara-Mahaica, Guyana